CLINICAL TRIAL: NCT00724113
Title: Evaluation of the Effectiveness of ARTHRO -Distension Plus Intensive Mobilisation in Shoulder Capsulitis
Brief Title: ARTHRO Distension Plus Intensive Mobilisation in Shoulder Capsulitis
Acronym: CAPSULITE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P051039
Record Dates: First submitted 2008-04-09; First posted 2008-07-29 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2014-05

CONDITIONS: Shoulder Capsulitis
Keywords: Shoulder capsulitis; ARTHRO distension; Mobilisation; Randomised clinical trial

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): infiltration intra articular
  Interventions: Procedure: infiltration intra articular
- 2 (Experimental): ARTHRO distension plus intensive mobilisation
  Interventions: Procedure: ARTHRO distension plus intensive mobilisation

INTERVENTIONS:
Procedure: infiltration intra articular — infiltration intra articular at inclusion with XYLOCAINE 1%
  Other Names: infiltration intra articular at inclusion with XYLOCAINE 1%
  Arms: 1
Procedure: ARTHRO distension plus intensive mobilisation — ARTHRO distension plus intensive mobilisation
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the effectiveness of ARTHRO distension plus intensive mobilisation in shoulder capsulitis.

DETAILED DESCRIPTION:
The aim of the study is to evaluate a treatment of shoulder capsulitis that associates ARTHRO distension and intensive mobilisation at 2, 6, 12, 26 and 52 weeks. It is a bicentric 87-month (inclusion: 74 months; follow up: 13 months) observer blind randomised clinical trial using 2 groups in parallel. The number of patients to be included is 66. The treatment that is evaluated associates ARTHRO distension followed by mobilisation of the shoulder 6 hours per day during 5 days, and then sessions of physiotherapy for 4 weeks. The control intervention is one intra-articular injection of corticosteroids and physiotherapy. The primary outcome is SPADI, namely pain and disability, at 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* shoulder capsulitis
* duration of symptoms ≥ 3 months
* health insurance

Exclusion Criteria:

* cognitive disorders
* Hypo coagulation
* biological inflammatory syndrome
* uncontrolled diabetes
* XYLOCAINE allergy
* pregnancy
* unable to understand and to speak french
* previous surgery of shoulder
* shoulder infiltration or distension in the previous month
* local contraindication to shoulder infiltration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-02; Primary Completion 2013-08 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pain and disability using SPADI score at 2 weeks | at 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johann Beaudreuil, PH MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Rheumatology department of Lariboisiere hospital, Paris, France

REFERENCES:
- [Derived] Jacob L, Lasbleiz S, Sanchez K, Morchoisne O, Lefevre-Colau MM, Nguyen C, Rannou F, Feydy A, Portal JJ, Schnitzler A, Vicaut E, Laredo JD, Richette P, Orcel P, Beaudreuil J. Arthro-distension with early and intensive mobilization for shoulder adhesive capsulitis: A randomized controlled trial. Ann Phys Rehabil Med. 2024 Sep;67(6):101852. doi: 10.1016/j.rehab.2024.101852. Epub 2024 Jun 1. PMID 38824872